CLINICAL TRIAL: NCT07015060
Title: Pathogenic Mechanisms Involved in the Initiation and Progression of Systemic Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PathSSC
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Scleroderma (Limited and Diffuse)
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PathSSc (Other)
  Interventions: Procedure: cutaneous biospy

INTERVENTIONS:
Procedure: cutaneous biospy — cutaneous biospy

SUMMARY:
Identify rare variants in candidate genes and pathways identified in familial SSc, in patients with sporadic SSc.

Perform (spatial) transcriptomic and proteomic analyses of affected skin from patients with and without cutaneous fibrosis, for the patterns and levels of expression/activation of candidate genes and pathways.

Test for dysregulation of expression/activation of candidate genes and pathways in live cells isolated from the blood and skin biopsy of patients, and for the impact of these dysregulations on cell appearance, behavior and function.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with one of the following:

  * Limited SSc
  * Limited cutaneous SSc
  * Diffuse cutaneous SSc
* Patients followed regularly in consultations at CUSL.
* Patients between ages 18-80.

Exclusion Criteria:

* Other (co-occurring) autoimmune/autoinflammatory disease
* Pregnancy
* Participants with temporary or definitive disabilities to give consent
* Participants unable to sign or read the inform consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Identify rare variants in candidate genes and pathways in SSC patients (blood and skin biopsy) | Through the entire study, approximately during 5 years
  Genetic analyses in affected skin from patients (Next Generation sequencing, (single cell) RNASeq, real time qPCR)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Limaye, PhD, Study Director — Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No